CLINICAL TRIAL: NCT02570854
Title: A First-in-human, Two-part (Open Label, and Randomized/Double Blind/Placebo Controlled), Single- and Repeat-dose Study of CSJ137 in Erythropoietin-treated Chronic Hemodialysis Patients With Functional Iron-deficiency Anemia
Brief Title: A Two-part Single- and Repeat-dose Study of CSJ137 in Anemic Chronic Hemodialysis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCSJ137X2201; 2017-002926-19 (EudraCT Number)
Record Dates: First submitted 2015-09-29; First posted 2015-10-07 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Anemia, Iron-Deficiency
Keywords: Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSJ137 (Experimental): In Part 1 up to 48 subjects will receive a single dose of CSJ137. In Part 2, up to 40 patients will be randomized to one of 2 arms with equal allocation: one CSJ137 dose arm from Part 1 and a placebo arm. Each patient in Part 2 will receive up to 2 doses (repeat dose).
  Interventions: Biological: CSJ137
- Placebo (Placebo Comparator): In Part 2, up to 40 patients will be randomized to one of 2 arms with equal allocation: one CSJ137 dose arm from Part 1 and a placebo arm. Each patient in Part 2 will receive up to 2 doses (repeat dose).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CSJ137 — Starting dose is 0.010 mg/kg and dose escalation will proceed with semi-log increase steps to a maximum dose level 10 mg/kg. Subjects receive the treatment via up to 30 minutes intravenous infusion.
  Arms: CSJ137
Drug: Placebo — Subjects will be dosed with a matching placebo (vehicle control) via up to 30 minutes intravenous infusion.
  Arms: Placebo

SUMMARY:
The study will assess the safety, tolerability and efficacy of CSJ137 in chronic hemodialysis patients. It is hypothesized that treatment with CSJ137 may improve the level of hemoglobin in patients on chronic hemodialysis with iron-restricted anemia while reducing the need for dosing with erythropoietin and intravenous iron in these patients.

DETAILED DESCRIPTION:
This posting discloses information about Part 1 of CCSJ137X2201. Another part, Part 2, of this trial was planned for conduct subsequent to the initiation of Part 1 and would have a different design than Part 1. However, due to internal strategic non-safety related decision, Part 2 is not going to be conducted and the trial will be terminated after Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodialysis-dependent for at least 2 months prior to screening.
2. Receiving hemodialysis at least 2 times per week
3. Receiving erythropoietin (EPO) therapy.
4. Hemoglobin (Hgb) ≥ 8.5 and < 11.5 g/dL at screening.
5. Ferritin >500 ng/mL and ≤ 2000 ng/mL at screening.
6. TSAT ≤ 50% at a minimum of one time point during the 90 days prior to baseline.

Exclusion Criteria:

1. Known diagnosis of hemochromatosis, bone marrow malignancy, lymphatic malignancy or myelodysplastic syndrome.
2. History of dialysis AV fistula thrombosis within 2 months prior to screening, or 2 or more episodes of AV fistula thrombosis within 6 months prior to screening.
3. Liver disease/dysfunction (Child-Pugh score ≥ 6), prior liver transplant, heart failure (NYHA Class III or IV); gastrointestinal bleeding.
4. A positive Hepatitis B surface antigen test result. Patients with Hepatitis C Virus (HCV) infection may be included if all other liver function eligibility criteria are met.
5. ALT, AST or bilirubin ≥ 1.5x ULN within 4 weeks prior to baseline.
6. Uncontrolled renal osteodystrophy
7. Conditions predisposing to an increased risk of serious infection, such as an indwelling vascular catheter (central venous line or non-tunneled/acute hemodialysis catheter) or active infection requiring antibiotic therapy at any time during the 2 weeks prior to screening. Tunneled hemodialysis catheters, and other "permanent" catheters are permitted.
8. Blood transfusion administered within 4 weeks prior to baseline.
9. Patients who received CSJ137 dose in the past.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | baseline through 115 days after CSJ137 is administered
  safety and tolerability following administration of CSJ137
Minimum active dose of CSJ137 determined by assessment of levels of hemoglobin in blood, without evidence of liver dysfunction or other safety concerns. | Hemoglobin response at 28 days post-dose
  to determine the minimum dose of CSJ137 that is active for treatment

SECONDARY OUTCOMES:
Peak concentration (Cmax) of CSJ137 in serum | before CSJ137 is administered, then 0.5 hours and 6 hours after CSJ137 is administered on Day 1. Also 1, 2, 3, 5, 12, 19, 28, and 84 days after CSJ137 is administered
  to assess the concentration of CSJ137 in the body over time
Area under the serum concentration versus time curve (AUC) | before CSJ137 is administered, then 0.5 hours and 6 hours after CSJ137 is administered on Day 1. Also 1, 2, 3, 5, 12, 19, 28, and 84 days after CSJ137 is administered
  to assess the concentration of CSJ137 in the body over time

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Lakewood, Colorado
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Chattanooga, Tennessee
- Novartis Investigative Site, Prague, Czechia
- Israel (6):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Hadera
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Results for CCSJ137X2201 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17809
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=712